CLINICAL TRIAL: NCT01063972
Title: Centralized Disease Management for Rural Hospitalized Smokers
Brief Title: Smoking Cessation in Rural Hospitals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Ellerbeck, MD, MPH (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Edward Ellerbeck, MD, MPH, Professor, Chairman Preventive Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01CA101963-07 (NIH); 5R01CA101963-07 (NIH)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental 1 (Experimental): Experimental: 1 Centralized disease management
  Interventions: Behavioral: Centralized disease management (CDM)
- Experimental 2 (Experimental): Experimental: 2 Counseling alone
  Interventions: Behavioral: Counseling (C)

INTERVENTIONS:
Behavioral: Centralized disease management (CDM) — Centralized Disease Management (CDM) arm will receive smoking cessation counseling with coordination of pharmacotherapy with their insurance coverage and their health care provider
  Arms: Experimental 1
Behavioral: Counseling (C) — Counseling (C) arm will receive counseling without the care coordination services.
  Arms: Experimental 2

SUMMARY:
Our long-term goal is to improve smoking cessation treatment for rural smokers. The objective is to assess the effectiveness of a centralized disease management program for hospitalized smokers that coordinates care across treatment settings and links smokers to existing resources. Our central hypothesis is that Centralized Disease Management (CDM) will increase the use of smoking cessation treatments and lead to greater long term smoking cessation than Counseling alone. Demonstrating the effectiveness of a disease management program and identifying the critical components of such a program will provide a basis for improving the utilization of existing smoking cessation resources while enhancing the treatment of rural hospitalized smokers.

DETAILED DESCRIPTION:
The proposed study will use a randomized clinical trial design to examine the effectiveness of centralized disease management (CDM) versus counseling alone (C) for smoking cessation. Hospitalized smokers in 30 rural critical access hospitals will be randomly assigned to either CDM (n=303) or C (n=303). Participants in both arms of the study will receive in-hospital smoking cessation counseling via telephone followed by 4 outpatient telephone-based counseling calls. The content and timing of these counseling calls are designed to emulate models of smoking cessation counseling that have been previously shown to be effective for hospitalized smokers. For recipients assigned to CDM, the counseling will be streamlined to allow time on the calls for specific disease management interventions, including screening for contraindications to pharmacotherapy and linking medication choices to the smoker's insurance coverage. After completing calls with CDM participants, the Tobacco Treatment Specialists will coordinate therapy with the patient's health care providers by providing them with brief consultation reports, prepared order sheets for inpatient treatment, and outpatient prescription requests. Six months postdischarge, participants in both groups will be contacted again, and persistent or relapsed smokers will be offered another cycle of the C or CDM intervention.

Assessments will be conducted at baseline and at months 3, 6, and 12. The primary outcome of interest will be biochemically verified 7-day point prevalence abstinence at 12 months. Secondary endpoints include number of quit attempts and number of cigarettes smoked (among continuing smokers), pharmacotherapy utilization, duration of pharmacotherapy utilization, and the extent of discussions with the healthcare provider. We will also examine the marginal cost-effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in a participating rural hospital
* Aged 18 years or older
* Smoke cigarettes on >25 of the last 30 days
* Have a home address and telephone
* Willing to participate in phone assessments

Exclusion Criteria:

* Terminal medical condition with life expectancy <1 year
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2010-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Ellerbeck, MD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Ellerbeck EF, Cox LS, Hui SA, Keighley J, Hutcheson TD, Fitzgerald SA, Cupertino AP, Greiner KA, Rigotti NA, Miller NH, Rabius V, Richter KP. Impact of Adding Telephone-Based Care Coordination to Standard Telephone-Based Smoking Cessation Counseling Post-hospital Discharge: a Randomized Controlled Trial. J Gen Intern Med. 2019 Dec;34(12):2804-2811. doi: 10.1007/s11606-019-05220-2. Epub 2019 Jul 31. PMID 31367875

RESULTS

PARTICIPANT FLOW:
Groups:
- Centralized Disease Management (CDM): Experimental: 1 Centralized disease management
  Centralized disease management (CDM): Centralized Disease Management (CDM) arm will receive smoking cessation counseling with coordination of pharmacotherapy with their insurance coverage and their health care provider
- Counseling (C): Experimental: 2 Counseling alone
  Counseling (C): Counseling (C) arm will receive counseling without the care coordination services.
Period: Overall Study
Arm/Group | Centralized Disease Management (CDM) | Counseling (C)
Started | 310 | 296
Completed | 296 (Participants who were deceased or incarcerated were excluded.) | 284 (Participants who were deceased or incarcerated were excluded.)
Not Completed | 14 | 12
Not completed — Death | 12 | 11
Not completed — Incarcerated | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Centralized Disease Management (CDM) | Counseling (C) | Total
Number analyzed (Participants) | 310 | 296 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (12.89) | 51.0 (11.82) | 50.8 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 189 | 383
  Male | 116 | 107 | 223
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 9 | 34
  Not Hispanic or Latino | 285 | 287 | 572
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 12 | 24
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 12 | 26
  White | 278 | 270 | 548
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 310 | 296 | 606
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes/day] | 19.3 (9.99) | 19.7 (10.84) | 19.4 (10.41)
Smokes within 30 minutes of waking [Count of Participants; unit: Participants] | 257 | 244 | 501
Fagerstrom score (heavy nicotine dependence) [Count of Participants; unit: Participants] — The modified Fagerström test score for nicotine dependence ranges from 0 to 6. Scores of 4 or higher indicate heavy smoking dependence
  Participants | 142 | 168 | 310
Motivation to quit smoking [Mean (Standard Deviation); unit: units on a scale] — Motivation to quit smoking scores range from 0 to 10, with 10 indicating high motivation.
  units on a scale | 9.3 (1.34) | 9.2 (1.60) | 9.3 (1.47)
Confidence to quit smoking [Mean (Standard Deviation); unit: units on a scale] — Confidence to quit smoking scores range from 0 to 10, with 10 indicating high confidence.
  units on a scale | 7.1 (2.61) | 6.8 (2.45) | 7.0 (2.53)
Planning to quit smoking in the next 30 days [Count of Participants; unit: Participants] | 303 | 285 | 588
Quit attempted in the past 6 months [Count of Participants; unit: Participants] | 169 | 154 | 323
Previous use of quit smoking medication [Count of Participants; unit: Participants] | 192 | 199 | 391

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 7-day Point Prevalence Abstinence From Cigarettes, Validated
Description: Participant-reported 7-day point prevalence abstinence from cigarettes, validated by salivary cotinine (< 15ng/ml) or proxy. Participants who did not respond to the survey were considered current smokers.
Time Frame: 12 months
Population: Participants who were deceased or incarcerated at month 12 were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Centralized Disease Management (CDM) | Counseling (C)
Number analyzed (Participants) | 296 | 284
Participants | 57 | 48
Statistical Analysis 1: Comparison: Centralized Disease Management (CDM) vs Counseling (C); Test type: Superiority; p = 0.46, Chi-squared

2. Secondary Outcome: Number of Participants With 7-day Point Prevalence Abstinence at 3 Months, Self-reported
Description: 7-day point prevalence abstinence at 3 months, self-reported. Participants who did not respond were considered smokers.
Time Frame: 3 months
Population: Participants who were deceased or incarcerated at month 3 were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Centralized Disease Management (CDM) | Counseling (C)
Number analyzed (Participants) | 303 | 292
Participants | 86 | 70
Statistical Analysis 1: Comparison: Centralized Disease Management (CDM) vs Counseling (C); Test type: Superiority; p = 0.22, Chi-squared

3. Secondary Outcome: Number of Participants With 7-day Point Prevalence Abstinence at 6 Months, Self-reported
Description: 7-day point prevalence abstinence at 6 months, self-reported. Participants who did not respond were considered smokers.
Time Frame: 6 months
Population: Participants who were deceased or incarcerated at month 6 were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Centralized Disease Management (CDM) | Counseling (C)
Number analyzed (Participants) | 301 | 290
Participants | 64 | 56
Statistical Analysis 1: Comparison: Centralized Disease Management (CDM) vs Counseling (C); Test type: Superiority; p = 0.56, Chi-squared

4. Secondary Outcome: Number of Participants With 7-day Point Prevalence Abstinence at 12 Months, Self-reported
Description: 7-day point prevalence abstinence at 12 months, self-reported. Participants who did not respond were considered smokers.
Time Frame: 12 months
Population: Participants who were deceased or incarcerated at month 6 were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Centralized Disease Management (CDM) | Counseling (C)
Number analyzed (Participants) | 296 | 284
Participants | 73 | 63
Statistical Analysis 1: Comparison: Centralized Disease Management (CDM) vs Counseling (C); Test type: Superiority; p = 0.48, Chi-squared

5. Secondary Outcome: Number of Participants Reporting Utilization of Smoking Cessation Pharmacotherapy During First 6 Months
Time Frame: 6 months
Population: Excludes participants who were deceased or incarcerated at month 6, or who did not report on pharmacotherapy use.
Measure: Count of Participants; unit: Participants
Arm/Group | Centralized Disease Management (CDM) | Counseling (C)
Number analyzed (Participants) | 264 | 254
Participants
  Any medication | 145 | 141
  Nicotine replacement therapy | 106 | 112
  Prescription medication | 58 | 45

6. Secondary Outcome: Number of Participants Reporting Utilization of Smoking Cessation Pharmacotherapy Between 6 and 12 Months
Time Frame: 12 months
Population: Includes only participants eligible to enter into Cycle 2 counseling (those who reported smoking at month 6). Excludes participants who were deceased or incarcerated at month 12, or who did not report on pharmacotherapy use.
Measure: Count of Participants; unit: Participants
Arm/Group | Centralized Disease Management (CDM) | Counseling (C)
Number analyzed (Participants) | 153 | 161
Participants
  Any medication | 80 | 68
  Nicotine replacement therapy | 50 | 50
  Prescription medication | 46 | 30

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Centralized Disease Management (CDM) | Counseling (C)
All-Cause Mortality (participants affected / at risk) | 12/310 | 11/296
Serious Adverse Events (participants affected / at risk) | 1/310 | 1/296
Other Adverse Events (participants affected / at risk) | 5/310 | 7/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Centralized Disease Management (CDM) (N=310) | Counseling (C) (N=296)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Centralized Disease Management (CDM) (N=310) | Counseling (C) (N=296)
Oral discomfort (Product Issues) | 1 (1) | 0 (0) — Tingling and blister associated with nicotine gum use
Dizziness (Product Issues) | 1 (1) | 1 (1)
Change in affect (Product Issues) | 2 (2) | 1 (1)
Sleep disturbance (Product Issues) | 1 (1) | 1 (1)
Headache (Product Issues) | 1 (1) | 1 (1)
Nausea (Product Issues) | 1 (1) | 1 (1)
Tremors (Product Issues) | 0 (0) | 1 (1)
Lightheadedness (Product Issues) | 0 (0) | 1 (1)
Local skin reaction (Product Issues) | 1 (1) | 0 (0) — Itching or rash at nicotine patch site
Loss of bladder control (Renal and urinary disorders) | 0 (0) | 1 (1) — One time, for a few moments
Constipation (Product Issues) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No